CLINICAL TRIAL: NCT02118441
Title: A Comparison of Ultrasound-Guided Versus Direct Palpation For Radial Artery Catheterization Among Cardiac Anesthesiologists
Brief Title: Ultrasound-guided Versus Direct Palpation Radial Artery Catheter Insertion Among Cardiac Anesthesiologists
Acronym: art-line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H13-00494
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Time to Insertion of Radial Artery Cannulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- direct palpation (Active Comparator): Radial artery catheter insertion will be conducted by direct palpation and use of anatomic knowledge by the Anesthesiologist.
  Interventions: Device: Direct Palpation-guided Radial Artery Catheter insertion
- Ultrasound (Active Comparator): Radial artery catheter insertion will be conducted by ultrasound guidance. A Sono-site ilook 25 Ultrasound (Sono-site, Inc., Bothell, WA, USA) with a 10-5 MHz linear array ultrasound transducer will be used.
  At the discretion on the Anesthesiologist, an out-of-plane (i.e. needle plane at right angles to ultrasound plane) will be used. Colour flow doppler may also be used to identify the artery if necessary.
  Interventions: Device: Ultrasound-guided Radial Artery Catheter Insertion

INTERVENTIONS:
Device: Ultrasound-guided Radial Artery Catheter Insertion
  Arms: Ultrasound
Device: Direct Palpation-guided Radial Artery Catheter insertion
  Arms: direct palpation

SUMMARY:
When a patient undergoes heart surgery, their Anesthesiologist will insert a tiny plastic tube, called a catheter, in the artery of the patient's wrist. This is called a radial artery catheter. A radial artery catheter allows accurate measurement of the patient's blood pressure during surgery. There are two common techniques for placing the radial artery catheter. The first is a "blind" technique whereby the Anesthesiologist feels for the pulse in the patient's wrist and places the catheter using the location of the pulse as a guide. The second technique, less commonly used, is one whereby the Anesthesiologist uses an ultrasound machine (painless to the patient) to "see" the artery, and thereby uses the ultrasound to guide the catheter placement. Our study will test the hypothesis that ultrasound-guided radial artery catheterization will have faster insertion times, with fewer complications compared with palpation-guided insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery
* Age 19 or older
* Provided written informed consent

Exclusion Criteria:

* Suspected inability to comply with study procedures, including language difficulties or medical history and/or concomitant disease, as judged by the investigator
* Previous surgery at the site of proposed radial artery catheterization
* Any vascular condition that may preclude eligibility for radial artery line insertion as judged by the investigator
* Patients with ventricular assist devices
* Previous inclusion in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Head, MD, Principal Investigator — Providence Health & Services
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140
- [Derived] Peters C, Schwarz SK, Yarnold CH, Kojic K, Kojic S, Head SJ. Ultrasound guidance versus direct palpation for radial artery catheterization by expert operators: a randomized trial among Canadian cardiac anesthesiologists. Can J Anaesth. 2015 Nov;62(11):1161-8. doi: 10.1007/s12630-015-0426-8. Epub 2015 Jul 10. PMID 26159436

RESULTS

PARTICIPANT FLOW:
Groups:
- Direct Palpation: Radial artery catheter insertion was conducted by direct palpation and use of anatomic knowledge by the Anesthesiologist.
  Direct Palpation-guided Radial Artery Catheter insertion
- Ultrasound: Radial artery catheter insertion was conducted by ultrasound guidance. A Sono-site ilook 25 Ultrasound (Sono-site, Inc., Bothell, WA, USA) with a 10-5 MHz linear array ultrasound transducer was used.
  At the discretion on the Anesthesiologist, an out-of-plane (i.e. needle plane at right angles to ultrasound plane) was used. Colour flow doppler may have also been used to identify the artery if necessary.
  Ultrasound-guided Radial Artery Catheter Insertion
Period: Overall Study
Arm/Group | Direct Palpation | Ultrasound
Started | 65 | 64
Completed | 62 | 63
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Direct Palpation: Radial artery catheter insertion will be conducted by direct palpation and use of anatomic knowledge by the Anesthesiologist.
  Direct Palpation-guided Radial Artery Catheter insertion
- Ultrasound: Radial artery catheter insertion will be conducted by ultrasound guidance. A Sono-site ilook 25 Ultrasound (Sono-site, Inc., Bothell, WA, USA) with a 10-5 MHz linear array ultrasound transducer will be used.
  At the discretion on the Anesthesiologist, an out-of-plane (i.e. needle plane at right angles to ultrasound plane) will be used. Colour flow doppler may also be used to identify the artery if necessary.
  Ultrasound-guided Radial Artery Catheter Insertion
- Total: Total of all reporting groups
Arm/Group | Direct Palpation | Ultrasound | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (14) | 67 (14) | 67 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 46 | 52 | 98
Region of Enrollment [Number; unit: participants]
  Canada | 62 | 63 | 125
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27 (5) | 26 (4) | 26.5 (4.5)
ASA physical status IV [Number; unit: participants] — American Society of Anesthesiologists (ASA) status is a system for assessing fitness for surgery. Class IV refers to patients who have severe systemic disease that is a constant threat to life. Status I refers to a healthy patient. Status II refers to patients with mild systemic disease. Status III refers to patients who have severe systemic disease. Thus ASA class IV patients are associated with higher morbidity and mortality compared to ASA 1 patients.
  participants | 61 | 59 | 120
Peripheral vascular disease [Number; unit: participants] | 3 | 3 | 6
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 140 (18) | 140 (21) | 140 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Time to Successful Radial Arterial Catheterization
Description: The time to successful radial arterial catheterization was defined as time zero to time of placement. Time zero for the DP group began when the anesthesiologist's fingers were placed on the patient with the purpose of palpating the artery. Time zero for the US group began when the US transducer was first placed on the patient's skin for the purpose of identifying the radial artery. Time to placement was defined as the interval from time zero until the time at which an arterial tracing was viewed on the monitor.
Time Frame: up to 5 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Direct Palpation | Ultrasound
Number analyzed (Participants) | 62 | 63
seconds | 104 [76 to 212] | 104 [68 to 270]

2. Secondary Outcome: Number of Attempts
Description: An attempt was defined as a new purposeful penetration of the skin with the needle (i.e., following complete withdrawal of the needle from the skin).
Time Frame: up to 5 minutes
Measure: Median (Inter-Quartile Range); unit: number of attempts
Arm/Group | Direct Palpation | Ultrasound
Number analyzed (Participants) | 62 | 63
number of attempts | 1 [1 to 2] | 1 [1 to 2]

3. Secondary Outcome: Number of Re-directions
Description: A re-direct was defined as the needle being purposefully withdrawn at least 5 mm and re-directed (but not removed from the skin entirely).
Time Frame: up to 5 minutes
Measure: Median (Inter-Quartile Range); unit: number of re-directs
Arm/Group | Direct Palpation | Ultrasound
Number analyzed (Participants) | 62 | 63
number of re-directs | 2 [0 to 6] | 3 [1 to 5]

4. Secondary Outcome: Complication Rate (Hematoma)
Description: A hematoma was defined a collection of blood or formation of a bruise surrounding the site of radial artery catheterization
Time Frame: up to 5 minutes
Measure: Number; unit: percentage of participants
Groups:
- Ultrasound: Radial artery catheter insertion was conducted by ultrasound guidance. A Sono-site ilook 25 Ultrasound (Sono-site, Inc., Bothell, WA, USA) with a 10-5 MHz linear array ultrasound transducer was used.
  At the discretion on the Anesthesiologist, an out-of-plane (i.e. needle plane at right angles to ultrasound plane) was used. Colour flow doppler may also have been used to identify the artery if necessary.
  Ultrasound-guided Radial Artery Catheter Insertion
Arm/Group | Direct Palpation | Ultrasound
Number analyzed (Participants) | 62 | 63
percentage of participants | 22.6 | 11.1

ADVERSE EVENTS:
Arm/Group | Direct Palpation | Ultrasound
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 14/62 | 7/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct Palpation (N=62) | Ultrasound (N=63)
hematoma (Vascular disorders) | 14 (14) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No